CLINICAL TRIAL: NCT02951702
Title: Oral Vancomyin for Primary Clostridium Difficile Infection Prophylaxis in Patients Receiving High-Risk Antibiotics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Luke's Hospital, Chesterfield, Missouri (Other)
Responsible Party: Principal Investigator, Ryan Medas, PGY2 Pharmacy Internal Medicine Resident, St. Luke's Hospital, Chesterfield, Missouri
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 940920-2
Record Dates: First submitted 2016-10-30; First posted 2016-11-01 (Estimated); Results first posted 2017-12-27 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-11

CONDITIONS: Clostridium Difficile Infection; Prophylaxis; Vancomycin
MeSH Terms: conditions — Clostridium Infections | interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): This will be the historical arm that has not received oral vancomycin but match criteria for "high risk"
- Vancomycin Oral (Experimental): This arm will receive oral vancomycin 125 mg daily if "high risk" and determined to be appropriate by an ID physician Intervention type: drug, vancomycin 125 mg daily
  Interventions: Drug: Vancomycin Oral

INTERVENTIONS:
Drug: Vancomycin Oral — This arm will receive oral vancomycin 125 mg daily if "high risk" and determined to be appropriate by an ID physician
  Other Names: Oral vancomycin; vancomycin
  Arms: Vancomycin Oral

SUMMARY:
The purpose of this study is to determine if oral vancomycin used as primary Clostridium difficile prophylaxis can reduce the incidence of this infection in high-risk patients.

DETAILED DESCRIPTION:
Clostridium difficile infection is a common healthcare-associated infection and one that is associated with significant morbidity as well as a risk for mortality. Current practice throughout the United States is targeted at infection prevention measures such as hand washing and isolation. Despite these measures, incidence of Clostridium difficile infections continue to rise as some institutions, including our own. Recently, a study published in Clinical Infectious Diseases found oral vancomycin for secondary prophylaxis to reduce the incidence of recurrence. No studies to date have evaluated primary prophylaxis with oral vancomycin. This will be a single center, prospective study to evaluate oral vancomycin use as primary Clostridium difficile prophylaxis. Patients treated by infectious disease physicians will be identified as "high risk" and after pager notification the ID physician will have the option to start oral vancomycin 125 mg by mouth daily if they determine it to be appropriate. Risk factors include age older than 65 years, taking gastric acid suppression medication, and receiving select broad-spectrum antibiotics. Oral vancomycin will be continued until de-escalation of antibiotics or hospital discharge and patients will be evaluated for Clostridium difficile infection development from the current hospital admission up to 4 weeks following antibiotic discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* "High-risk" patients defined as: age older than 65, on gastric acid suppression, and select antibiotics
* Gastric acid suppression includes proton pump inhibitors and histamine-2 receptor antagonists
* Selected antibiotics include fluoroquinolone (ciprofloxacin, levofloxacin), clindamycin, a 3rd or 4th generation cephalosporin, a broad-spectrum aminopenicillin (ampicillin-sulbactam, piperacillin-tazobactam), or a carbapenem

Exclusion Criteria:

* Failure to meet all three requirements for "high risk"
* Vancomycin allergy
* Active clostridium difficile infection prior to inclusion
* Prophylactic oral vancomycin prior to study inclusion (i.e. prolonged vancomycin taper)
* Receipt of medications that also treat Clostridium difficile (metronidazole, rifaximin, fidaxomicin)
* Pregnant or breastfeeding

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-11; Primary Completion 2017-05 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan E Medas, PharmD, Principal Investigator — St. Luke's Hospital

REFERENCES:
- [Background] Lessa FC, Mu Y, Bamberg WM, Beldavs ZG, Dumyati GK, Dunn JR, Farley MM, Holzbauer SM, Meek JI, Phipps EC, Wilson LE, Winston LG, Cohen JA, Limbago BM, Fridkin SK, Gerding DN, McDonald LC. Burden of Clostridium difficile infection in the United States. N Engl J Med. 2015 Feb 26;372(9):825-34. doi: 10.1056/NEJMoa1408913. PMID 25714160
- [Background] O'Brien JA, Lahue BJ, Caro JJ, Davidson DM. The emerging infectious challenge of clostridium difficile-associated disease in Massachusetts hospitals: clinical and economic consequences. Infect Control Hosp Epidemiol. 2007 Nov;28(11):1219-27. doi: 10.1086/522676. Epub 2007 Oct 3. PMID 17926270
- [Background] Cohen SH, Gerding DN, Johnson S, Kelly CP, Loo VG, McDonald LC, Pepin J, Wilcox MH; Society for Healthcare Epidemiology of America; Infectious Diseases Society of America. Clinical practice guidelines for Clostridium difficile infection in adults: 2010 update by the society for healthcare epidemiology of America (SHEA) and the infectious diseases society of America (IDSA). Infect Control Hosp Epidemiol. 2010 May;31(5):431-55. doi: 10.1086/651706. PMID 20307191
- [Background] Owens RC Jr, Donskey CJ, Gaynes RP, Loo VG, Muto CA. Antimicrobial-associated risk factors for Clostridium difficile infection. Clin Infect Dis. 2008 Jan 15;46 Suppl 1:S19-31. doi: 10.1086/521859. PMID 18177218
- [Background] Magill SS, Edwards JR, Bamberg W, Beldavs ZG, Dumyati G, Kainer MA, Lynfield R, Maloney M, McAllister-Hollod L, Nadle J, Ray SM, Thompson DL, Wilson LE, Fridkin SK; Emerging Infections Program Healthcare-Associated Infections and Antimicrobial Use Prevalence Survey Team. Multistate point-prevalence survey of health care-associated infections. N Engl J Med. 2014 Mar 27;370(13):1198-208. doi: 10.1056/NEJMoa1306801. PMID 24670166
- [Background] Marra F, Ng K. Controversies Around Epidemiology, Diagnosis and Treatment of Clostridium difficile Infection. Drugs. 2015 Jul;75(10):1095-118. doi: 10.1007/s40265-015-0422-x. PMID 26113167
- [Background] Van Hise NW, Bryant AM, Hennessey EK, Crannage AJ, Khoury JA, Manian FA. Efficacy of Oral Vancomycin in Preventing Recurrent Clostridium difficile Infection in Patients Treated With Systemic Antimicrobial Agents. Clin Infect Dis. 2016 Sep 1;63(5):651-3. doi: 10.1093/cid/ciw401. Epub 2016 Jun 17. PMID 27318333
- [Background] Johnson S. Editorial Commentary: Potential Risks and Rewards With Prophylaxis for Clostridium difficile Infection. Clin Infect Dis. 2016 Sep 1;63(5):654-5. doi: 10.1093/cid/ciw424. Epub 2016 Jun 28. No abstract available. PMID 27358349

RESULTS

PARTICIPANT FLOW:
Groups:
- Vancomycin: This arm will receive oral vancomycin 125 mg daily if "high risk" and determined to be appropriate by an ID physician
  Vancomycin Oral: This arm will receive oral vancomycin 125 mg daily if "high risk" and determined to be appropriate by an ID physician
Period: Overall Study
Arm/Group | Control | Vancomycin
Started | 34 | 17
Completed | 34 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Vancomycin | Total
Number analyzed (Participants) | 34 | 17 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 34 | 17 | 51
Age, Continuous [Mean (Full Range); unit: years] | 76 [65 to 90] | 75 [65 to 86] | 75 [65 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 13 | 30
  Male | 17 | 4 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 34 | 17 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34 | 17 | 51

OUTCOME MEASURES:

1. Primary Outcome: Clostridium Difficile Infection Occurrence
Description: The incidence of clostridium difficile infection as detected for GDH/toxin positive or PCR if the GDH/toxin is equivocal.
Time Frame: Within 4 weeks from the completion of antibiotic treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Vancomycin
Number analyzed (Participants) | 34 | 17
Participants | 2 | 0

2. Secondary Outcome: Time to Clostridium Difficile Infection Occurence
Description: This is the time from the start of antibiotics to the diagnosis of clostridium difficile.
Time Frame: Within 4 weeks from completion of antibiotic treatment
Measure: Mean (Full Range); unit: days
Arm/Group | Control | Vancomycin
Number analyzed (Participants) | 34 | 17
days | 2 [0 to 2] | 0 [0 to 0]

3. Secondary Outcome: Clostridium Difficile Infection Severity
Description: Severity as defined by the IDSA/SHEA guidelines (mild to moderate, defined as white-cell count less than 15,000 cells/µL or increase in serum creatinine (SCr) by <1.5 times the baseline; severe, defined as white-cell count greater than 15,000 cells/µL or increase in SCr by >1.5 times the baseline; and fulminant, defined as the criteria above for severe with shock, hypotension, ileus, or megacolon)
Time Frame: Within 4 weeks from completion of antibiotic treatment
Measure: Number; unit: participants
Arm/Group | Control | Vancomycin
Number analyzed (Participants) | 34 | 17
participants
  Mild-Mod | 1 | 0
  Severe | 1 | 0

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Control | Vancomycin
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/17
Other Adverse Events (participants affected / at risk) | 0/34 | 0/17

LIMITATIONS AND CAVEATS:
Underpowered study; primary outcome relied upon patient's developing CDI while in the hospital or follow up at the study hospital.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-27): https://cdn.clinicaltrials.gov/large-docs/02/NCT02951702/Prot_SAP_000.pdf